CLINICAL TRIAL: NCT03144414
Title: Laparoscopic Assisted Doderlin Vaginal Hysterectomy vs. Laparoscopic Assisted Vaginal Hysterectomy: A Randomized Clinical Trial.
Brief Title: Laparoscopic Assisted Doderlin Vaginal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1393
Record Dates: First submitted 2017-04-30; First posted 2017-05-08 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Laparoscopic Hysterectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAVH (Active Comparator): Laparoscopic Assisted Vaginal Hysterectomy
  Interventions: Procedure: Laparoscopic hysterectomy
- LADH (Active Comparator): Laparoscopic Assisted Doderlin Vaginal Hysterectomy
  Interventions: Procedure: Laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic hysterectomy — Laparoscopic hysterectomy
  Other Names: Laparoscopic Assisted Hysterectomy

SUMMARY:
This prospective randomized clinical trial will be conducted in Ain Shams University Maternity Hospital during the period from May 2017 to December 2017. Group Ι: 30 patients will undergo conventional laparoscopic assisted vaginal hysterectomy (LAVH). Group ΙΙ: 30 patients will undergo laparoscopic assisted Doderlein vaginal hysterectomy (LADH)

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years.
* Uterine size ≤ 14weeks.
* Benign uterine pathology (Fibroid uterus, endometrial hyperplasia, DUB, uterine prolapse).
* No contraindication for laparoscopic surgery.

Exclusion Criteria:

* Gynecologic malignancy.
* Contraindications to laparoscopy like any medical condition worsened by pneumoperitoneum or the Trendelenburg position.
* Large abdominal hernia
* Large ovarian mass
* History of previous laparotomy finding extensive adhesions

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Operative time | 24 hours

SECONDARY OUTCOMES:
postoperative pain | 24 hours
  questionnaire using Visual Analogue scale
operative complications | 24 hours
Hospital stay | 24 hours
Blood loss | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt